CLINICAL TRIAL: NCT02203812
Title: The Effect of Probiotic Lozenge Administration on Gingivitis and on Mild & Moderate Periodontitis: A Randomized Controlled Clinical Trial.
Brief Title: Effect of Probiotic Lozenge on Gingivitis and Periodontitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CD Pharma India Pvt. Ltd. (Industry)
Collaborators: Government Dental College and Hospital, Vijayawada, Andra Pradesh, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIJ_GIN-PRO 01
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Mild and Moderate Chronic Periodontitis
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic Arm (Experimental): L. brevis CD2 Lozenges (4 lozenges per day - 1 lozenge in the morning, 1 lozenge in the afternoon and 2 lozenges in the night). Each lozenge contains at least 1 billion colony forming units of Lactobacillus brevis CD2.
  Interventions: Drug: Probiotic Arm
- Placebo Arm (Placebo Comparator): Placebo lozenges (4 lozenges per day - 1 lozenge in the morning, 1 lozenge in the afternoon and 2 lozenges in the night). The placebo lozenge contains all ingredients except the active constituent (probiotic, Lactobacillus brevis CD2).
  Interventions: Drug: Placebo Arm

INTERVENTIONS:
Drug: Probiotic Arm — Each Inersan lozenge contains at least 1 billion colony forming unit of Lactobacillus brevis CD2
  Arms: Probiotic Arm
Drug: Placebo Arm — Placebo lozenges contain all ingredients except the active constituent (probiotic, Lactobacillus brevis CD2)
  Arms: Placebo Arm

SUMMARY:
The oral cavity is mostly influenced by general health. The oral microbiota which is as complex as the gastro-intestinal or vaginal microbiota are considered to be difficult therapeutic targets. The effects of probiotics in different fields of health care have resulted recently in the introduction of probiotics for oral healthcare. Probiotics have been clinically proved effective in different fields of oral healthcare such as halitosis, oral candidiasis and tooth decay. They have also been inducted in the field of periodontal healthcare because of the current views on the etiology of plaque- related periodontal inflammation.

ELIGIBILITY:
Inclusion Criteria

* Patients with chronic mild to moderate periodontitis.
* Having Pocket depth > 4mm.
* Mean loss of attachment, evaluated by measuring the distance from cement-enamel junction to the bottom of the probing pocket > 4mm

Exclusion Criteria:

* Patients on probiotic supplements
* Patients who have allergy to lactose and fermented milk products
* Smokers
* Patients who are on antibiotic therapy or were on antibiotic therapy in the past 6 months
* Patients with advanced periodontal and/or periapical conditions which necessitate immediate treatment
* Patient suffering from any systemic illness
* Patients who are deemed to be un-cooperative

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Improvement in Clinical Periodontal Indices | 8 weeks
  Improvement in clinical periodontal indices, namely, Plaque Index (PI), Gingival Index (GI), Probing Pocket Depth (PPD), Bleeding on Probing (BOP)

SECONDARY OUTCOMES:
Improvement in Biochemical Indices | 8 weeks
  Changes in levels of Inflammatory markers, namely, Interleukin 1β, Matrix metalloproteinases-8 (MMP), Myeloperoxidase (MPO) and Calprotectin in Gingival Crevicular Fluid (GCF)

CONTACTS AND LOCATIONS:
Overall Officials: Surya Jyotsna Kiran Kanchumurthy, BDS, Principal Investigator — Government Dental College and Hospital, Vijayawada, Andhra Pradesh; Narendra Dev Jampani, MDS, Study Director — Government Dental College and Hospital, Vijayawada, Andhra Pradesh; Vajra Madhuri S, MDS, Principal Investigator — Government Dental College and Hospital, Vijayawada, Andhra Pradesh
Locations (1):
- Department of Periodontology, Government Dental College & Hospital, Vijayawada, Andhra Pradesh, India